CLINICAL TRIAL: NCT02615834
Title: Testing the Ability of Gentle Chest Pressure to Maintain Peripheral Oxygenation in Intubated Pediatric Patients
Brief Title: Chest Pressure for Intubated Peds Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00060292
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Study group (Active Comparator)
  Interventions: Procedure: Gentle chest pressure

INTERVENTIONS:
Procedure: Gentle chest pressure — Gentle pressure on the patient's right chest will be applied to achieve 12 breaths per minute.
  Arms: Study group

SUMMARY:
We previously showed that a gentle chest pressure technique could be used on children over a year old to generate around 20% of the volume of air inhaled or exhaled in a single normal breath (also known as tidal volume). This showed that a non-invasive method could be used to provide a temporary means of artificial breathing, meaning that invasive procedures, such as putting in a breathing tube, could be avoided. What our results did not tell us, however, is how much oxygen can get to peripheral tissues (e.g., arms, legs) with this method. In this study, we want to compare two groups of children. All children will have a breathing tube; one group will have gentle chest pressure performed on them to see if oxygen saturations can be maintained above 90%. The other group will receive no chest pressure. We will see how long it takes for oxygen levels in both groups to drop to 90%, at which point, the patient will be ventilated mechanically.

DETAILED DESCRIPTION:
BACKGROUND Airway management is different in the pediatric population compared to adults mainly due to the differences in respiratory physiology and anatomy. The oxygen consumption is about three times as high in children than in adults resulting in a higher impact on oxygen delivery and reserve should there be a problem with ventilation in children. During inspiration, the vertical dimension of the chest cavity is increased and the rib margins are lifted and moved out, causing an increase in the transverse diameter of the thorax. This generates a negative pressure in the intrapleural space between the lungs and the chest wall resulting in lung inflation. The rib cages of young children are very pliable. One of the theoretical ways to improve the efficiency of lung inflation in small children with such compliant rib cage is to apply pressure on the chest. The intrathoracic pressure increases above atmospheric pressure and air preferentially flows out of the lungs according to the pressure gradient. When the pressure on the chest is released and the thorax recoils passively ("springs open"), a negative intrathoracic pressure is generated. This effectively "sucks" air into the lungs along the pressure gradient. Although age-related pliability differences may be present, we do not expect this to be a significant factor in using the chest pressure technique successfully.

We previously demonstrated that application of gentle pressure on the right chest of pediatric patients generated 20% of the tidal volume achieved with mechanical ventilation, regardless of whether the patient was intubated or not. Chest pressure was monitored using a force transducer and did not exceed the patient's body weight. Indeed, the pressure used was considerably less than what would be administered during cardiopulmonary resuscitation. There was little variation across age ranges; for each age group, we observed a difference of less than 1 mL/kg compared to the overall mean tidal volume. Our study also showed that the gentle chest pressure technique was well-tolerated by pediatric patients of any age (neonate to adolescent), and no adverse events were encountered, supporting this technique as a very low-risk maneuver.

While these results are encouraging, the study did not provide detailed information on how much peripheral oxygenation (SpO2) is achieved with the gentle chest pressure technique. An editorial that accompanied the published study supports further investigation of the technique, including the extent to which it provides ventilation and its ability to provide adequate oxygenation. In this study, we wish to perform the technique on pediatric patients to determine if it can be used to maintain SpO2 for a significant length of time. For safety purposes, all trials will be done on patients whose tracheae have been intubated.

OBJECTIVE To determine if a gentle chest pressure technique can be used to maintain SpO2 over 90% significantly longer than allowing SpO2 to desaturate spontaneously.

HYPOTHESIS Gentle chest pressure can maintain SpO2 over 90% for significantly longer than if tissues are allowed to desaturate spontaneously.

METHODS After obtaining ethics approval, informed consent with or without assent whenever is appropriate (usually above the age of 6 years) will be obtained on the day ward. Consent will be obtained by a research assistant not involved with the clinical care of the patient. The demographic details of the patients, such as age, weight, height, ASA and any medical conditions will be recorded. The patient will be taken into the operating room, and routine monitoring will be applied. After induction of a standard general anesthesia where the technique is at the discretion of each individual anesthesiologist responsible for the case, the patient's trachea will be intubated. The patient will be ventilated mechanically for two minutes to achieve 100% peripheral oxygen saturation.

During this time, the patient will be randomly allocated to one of two groups - intervention and control - by a member of the study team. Instructions in sealed envelopes will indicate whether the chest pressure technique will be used or not. For patients in the intervention group, the anesthesiologist will apply gentle pressure (not exceeding the patient's own weight) vertically down on the patient's right chest. In the previous study, we calibrated pressure using a force transducer; since then, the Stollery pediatric anesthesia staff has been employing the technique in regular practice and are well experienced with the amount of force needed to generate adequate tidal volume. Since a pre-defined distance to depress the chest (e.g., 1 or 2 cm) is difficult to use for a wide range of patients weights (approximately 9-67 kg range in the previous study), in this study, the anesthesiologist will apply pressure to the point where resistance is encountered and then release. Upon release of pressure, the anesthesiologist will wait for one second. In our experience, the time taken to apply downward pressure and allow for chest recoil lasts approximately four seconds which, with the one second pause following pressure release, creates a total time of 5 seconds for the entire maneuver. As such, the maneuver can be used to achieve 12 breaths per minute. Oxygen saturation will be monitored and recorded continuously. The time taken for SpO2 levels to fall to 90% will be recorded, at which point, the anesthesiologist will restart mechanical ventilation. If SpO2 values fall below 90% at any time while the chest pressure technique is being performed, the patient can be ventilated mechanically immediately because they are already intubated.

Patients randomized to the control group will receive the same care as the intervention group except that no chest pressure technique will be performed. Following mechanical ventilation to 100% SpO2, surgery will proceed as normal with no additional intervention (i.e., gentle chest pressure) by the anesthesiologist. Peripheral oxygen saturations will be monitored during this time, and once the level reaches 90%, the time will be recorded, and the anesthesiologist will restart mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients between one and 18 year of age
* Requirement for insertion of an endotracheal tube
* American Society of Anesthesiologists (ASA) class I to III

Exclusion Criteria:

* Failure to obtain parental consent or patient assent when appropriate (in general, children over 6 years of age)
* ASA IV
* Patients with any cardiac pathology
* Patients with any respiratory pathology
* Patients with any form of chest deformity, for example, pectus excavatum, pectus carinatum, scoliosis
* Patients who had previous cardiac or thoracic surgery

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Time for SpO2 level to reach 90% | Immediately following mechanical ventilation to 100% SpO2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Tsui BC, Horne S, Tsui J, Corry GN. Generation of tidal volume via gentle chest pressure in children over one year old. Resuscitation. 2015 Jul;92:148-53. doi: 10.1016/j.resuscitation.2015.02.021. Epub 2015 Mar 4. PMID 25749553
- [Background] Morgan RW, Nadkarni VM, Berg RA. Can gentle chest compressions result in substantial ventilation? Resuscitation. 2015 Jul;92:A2-3. doi: 10.1016/j.resuscitation.2015.04.003. Epub 2015 Apr 29. No abstract available. PMID 25936933